CLINICAL TRIAL: NCT06254105
Title: Feasibility of a Cross-sectorial Management Program in Hand Osteoarthritis
Acronym: HANDY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parker Research Institute (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Eva Ejlersen Wæhrens, Professor, Parker Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Parker Instituttet
Record Dates: First submitted 2024-01-22; First posted 2024-02-12 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hand Osteoarthritis
Keywords: Feasibility; Occupational therapy; Hand Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Cohort design involving people with hand OA, general practitioners and occupational therapist employing a mixed-method approach
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Receive the HANDY programme
  Interventions: Other: HANDY programme

INTERVENTIONS:
Other: HANDY programme — The manualised HANDY program includes descriptions of procedures related to the GP's evaluation of the client's need for referral to occupational therapy, procedures for referral from the GP to community-based occupational therapy, the group-based occupational therapy programme, and recommendations related to collaboration and communication between GP and occupational therapist.

SUMMARY:
To support the referral of people with Hand Osteoarthritis (HOA) to evidence-based occupational therapy addressing decreased ADL ability, a cross-sectorial management program for people with HOA, named HANDY, was developed. The HANDY program includes procedures for needs evaluation and referral, and a group-based occupational therapy program. The development was based on the United Kingdom's Medical Research Councils recommendations. A core element is involvement of stakeholders. Therefore, the research group has worked closely with GPs, OTs, people with HOA and specialist within rheumatology. Through a co-productional process the HANDY program was developed based on theories, research evidence, current best practice and the preferences of people with HOA. The aim of this study is to evaluate the feasibility of the HANDY

DETAILED DESCRIPTION:
Background Osteoarthritis (OA) occurs after the age of 40 and increases with age causing pain and stiffness mostly in knees, hands, and hips. Globally nearly 600 million people are affected and it is estimated to increase to 642 million in 2050 due to growth and ageing populations. Hand OA is the second most common OA subtype, and clinically hand OA can be seen with three clinically patterns, First were the distal and proximal interphalangeal joints are affected, secondly including the thumb base, or thirdly in a combination of the two before mentioned.

People with hand OA reports difficulties in relation to performance of Activities of Daily Living (ADL). More specifically, they report using extra time and/or effort and occasionally also need of help to manage daily life. ADL task performance problems may be in relation to personal ADL (PADL) tasks carried out every day such as bathing, dressing, and eating or instrumental ADL (IADL) tasks carried out on a weekly basis such as cleaning, cooking, and shopping. When people with hand OA are observed using standardized ADL assessment tool, the overall ADL motor ability also indicates clumsiness and use of extra effort for the population. When comparing the mean of ADL motor ability with other age-related healthy adults, people with hand OA have a lower ADL motor ability.

In 2020 OA was the top-ten leading cause of disability for older adults (>70 years). The increasing OA population presenting with decreased ADL ability will lead to a greater burden on the health care system. According to the 2018 EULAR recommendations, people with hand OA should be offered multidisciplinary and multimodal treatment approaches. In relation to non-pharmacological treatment education, training, home modifications, assistive devices, and splints to reduce symptoms and improve overall functioning and quality of life are recommended. Several of these treatment modalities may be employed by occupational therapists to improve ADL ability including education, home modifications, assistive devices, and splinting. Still, when exploring current practice of referring people with disabilities due to hand OA for occupational therapy among Danish general practitioners, only one were referred. Moreover, a literature review indicated a lack of an evidence-based occupational therapy program addressing decreased ADL ability among people with hand OA. Previous interventions studies involving people with hand OA have often focused on improving body functions (e.g. muscle strength) through exercises. This approach is based on the assumption that improved body function will lead to increased ability to perform ADL. Research, however, indicates that improved body function not necessarily translate into improved ADL ability. Rather, existing research support, that interventions focusing on ADL also has an effect on improvement of ADL ability for people with chronic condition.

To support the referral of people with hand OA to evidence-based occupational therapy addressing decreased ADL ability, a cross-sectorial management program for people with hand OA, named HANDY, was developed. The HANDY program includes procedures for needs evaluation and referral, and a group-based occupational therapy program. The development was based on the United Kingdom's Medical Research Councils recommendations. A core element is involvement of stakeholders. Therefore, the research group has worked closely with GPs, OTs, people with hand OA and specialist within rheumatology. Through a co-productional process the HANDY program was developed based on theories, research evidence, current best practice and the preferences of people with hand OA. The aim of this study is to evaluate the feasibility of the HANDY program.

Methods Aims The overall aim is to investigate the feasibility of the cross-sectorial management program, HANDY, for people with hand OA (v. 1.0) in terms of content and delivery of needs evaluation, referral procedures, the occupational therapy intervention, and the cross-sectorial collaboration.

More specifically, based on the guidance developed by O'Cathain:

1. Determine to what extent the HANDY program needs to be refined or adapted to make it more acceptable to users or more relevant or useful to the specific context in which it is delivered (Intervention development)?
2. Identify adjustments needed to improve relevance of the HANDY program for people with hand OA, general practitioners and occupational therapist, and determine which aspects are fixed and flexible (Intervention components)?
3. Determine which components that are meaningful and beneficial, and identify unintended positive/negative side effects (Perceived value, benefits, harms or unintended consequences).
4. Explore the overall perception of the content and delivery described in the HANDY program and if it is relevant to implement in practice (Acceptability in principle).
5. Explore to what extent people with hand OA, general practitioners and occupational therapist do think that the HANDY program can be implemented and if it varies across municipalities (Feasibility and acceptability in practice).
6. Determine the number of referrals in the HANDY program, as well as the number of sessions delivered for people with hand OA. Furthermore, the adherence to procedures described for the program, the duration of components in each session and if the dose was sufficient (Fidelity, reach and dose).

Aspects related to trial design and to development and refinement of program theory including mechanisms of actions will be explored in a future pilot-RCT study.

Design, settings This is a feasibility study using a cohort design involving people with hand OA, general practitioners and occupational therapist employing a mixed-method approach.

The feasibility of the HANDY program will be evaluated in two municipalities in the Capital Region of Denmark. The municipalities have approximately 48.000 and 56.000 inhabitants, respectively, and are both located near Copenhagen. In each municipality three general practitioners and one community-based rehabilitation centre will be involved. In one municipality the three general practitioners work in the same clinic, whereas in the other municipality they work in two different clinics. The rehabilitation centres are organised under the municipal health administration.

The occupational therapy part of the HANDY program will be delivered in the homes and in the rehabilitation centre. In the rehabilitation centre, sessions will be held in contextualized situations, where people with hand OA may be engaged in educational programs and practice strategies to improve ADL tasks performance. To ensure a representative sample and enough information about feasibility of the program, each municipality must complete two HANDY occupational therapy interventions.

Participants People diagnosed with hand OA (n=30), > 18 years and motivated to participate in a group program focusing on improvement in ADL task performance. General practitioners (GPs) (n=6) working in a clinic with agreement with the Danish health insurance receiving patients with all kinds of everyday symptoms and illnesses, who express interest in contributing to development and evaluation of a program for people with hand OA. Occupational therapists (OTs) (n=4) working with community-based rehabilitation and with six months of community-based working experience.

Recruitment

People with hand OA will be recruited by six GPs from January 5, 2024. When a person with hand OA consults the GP, the GP briefly informs about the research project (e.g., by saying: "this is a project offering a cross-sectorial management program, including a needs evaluation, and if relevant, referral for a group-based occupational therapy intervention addressing problems related to performance of daily activities related to hand OA"), and then asks if he/she is interested in learning more about the project. If the person confirms to be interested, the GP provides additional oral and written information on the project. If the person then confirms that he/she will participate, the GP obtains written consent as a prerequisite to initiate the HANDY program.

Cross-sectorial management program The first version of the HANDY program was developed based on the United Kingdom's Medical Research Councils recommendations. The manualised HANDY program includes descriptions of procedures related to the GP's evaluation of the client's need for referral to occupational therapy, procedures for referral from the GP to community-based occupational therapy, the group-based occupational therapy programme, and recommendations related to collaboration and communication between GP and occupational therapist.

* Needs evaluation The purpose of the needs evaluation is to clarify the relevance of referring the person with hand OA to community-based occupational therapy. The needs evaluation is conducted when a person with hand OA consults the GP with problems related to hand OA, or when problems related to hand OA are addressed during a consultation not related to hand OA in the first place. The needs evaluation is performed to determine if the hand OA affects the persons with hand OA daily life. First the GP asks questions related to how the person with hand OA perceives using the hands in performance of ADL tasks, e.g., zipping zippers when dressing, cutting nails, opening cans when cooking, or wringing a cloth when cleaning. Then a screening covering five aspects is conducted: 1) assessment of grip strength with, 2) assessment of problems turning things with the hands, for example turning a key in a lock, 3) assessment of problems related to turning up taps, 4) assessment of problems related to turning a round doorknob or handle, and 5) assessment of problems related to buttoning buttons. In step 1 hand strength is assessed by using simple handshake, and steps 2-5 are assessed asking the person with hand OA, and hence are based on self-report. All aspects are scored with yes or no. The person with hand OA is referred to community-based occupational therapy based on answering at least one of the questions with "yes".
* Referral procedures Referral is conducted using existing electronic procedures. As part of the referral the GP takes an anamnesis focusing on the persons with hand OA level of functioning and the identified problems related to daily life, including the specific diagnosis.

In the municipality the referral is received and processed according to standard procedures.

- Occupational Therapy program

The HANDY occupational therapy intervention follows the Occupational Therapy Intervention Process Model (OTIPM), specifying the steps of a problem-solving process focused on enabling participation in needed and important tasks in everyday life. The HANDY occupational therapy intervention consists of six mandatory sessions of 120 minutes. The intervention consists of a combination of individual and group sessions, with a maximum of eight people with hand OA in each group.

Session 1 consists of an individual session in the persons with hand OA home involving evaluations of self-reported and observed ADL task performance. The Activities of Daily Living Interview (ADL-I) is used to measure self-reported ADL ability, and the Assessment of Motor and Process Skills (AMPS) to measure observed ADL ability. Both ADL-I and AMPS are valid and reliable measurements for people with chronic conditions. Following the ADL evaluation, the person with hand OA and OT will together formulate goals for the intervention using the Goal Attainment Scale (GAS) and begin the speculations about reasons for decreased ADL ability.

Sessions 2 to 5 are group-based, held at the rehabilitations centre and involve peer learning activities. In session 2 the people with hand OA are introduced to how they can identify factors influencing their individual ADL task performances (using the Transactional Model of Occupation (TMO)) in plenum. The results of the individual analyses form the basis for sessions 3 to 5 focusing on improving ADL task performance by addressing these factors. The interventions are mainly based on compensatory strategies to improve ADL task, in relation to energy conservation (session 3), assistive devices and the use of orthoses (session 4). The last group sessions will also address how necessary and meaningful activities (e.g., ADL, leisure, or social activities) may be used to maintain hand function (session 5). The group sessions will be individualised based on the people with hand OA individual evaluation and problems with performing ADL tasks. The occupational therapy intervention is terminated with an individual session (session 6) in the person with hand OA home involving evaluation of goal attainment and changes in self-reported and observed ADL ability using ADL-I, AMPS and GAS.

- Communication and Collaboration After the final session of the occupational therapy intervention, the OT submits an epicrisis to the GP, including information on how the person with hand OA profited from the programme, any potential outcomes related to ADL ability, whether the person with hand OA was referred to other services in the municipality (e.g., physiotherapy or assistance in the home), and potential future recommendations.

Training of GPs and OTs To support that the HANDY program will be delivered according to the manual (fidelity), the GPs and OTs will be trained in procedures related to content and delivery. GPs will in a one-hour online session be trained in the procedures of needs evaluation, referral, and cross-sectorial collaboration. The OTs will participate in a two-day workshop with half day follow up before the first session of the occupational therapy intervention is delivered. They will be trained in the occupational therapy intervention, including evaluations of self-reported and observed ADL performance and procedures for goal setting, and in the cross-sectorial collaboration procedures.

Procedures for data collection:

A mixed-method approach will be used to gather data to explore aspects of content and delivery.

Registration forms will be collected during each step of the HANDY program in relation to research objectives 1 to 6. The GP fills out a registration form immediately after each consultation including a needs evaluation and when the overall program is finalised, i.e., when the GP receives an epicrisis from the occupational therapist. Moreover, the GP registrates the number of persons with hand OA declining the invitation to participate based on the initial information. OTs and people with hand OA will fill in registration forms after each intervention session.

Focus group interviews with people with hand OA will be carried out after completion of the occupational therapy program. Qualitative individual interviews with the GPs and qualitative focus group interviews with OTs will be conducted after the HANDY program has been completed. All interviews address research questions 1, 3, 4, and 5.

To determine change in ADL ability among people with hand OA, data in terms of ADL-I and AMPS will be collected at session 1 and 6 in the occupational therapy intervention. The ADL-I and the AMPS have demonstrated sensitivity to change among persons living with chronic conditions. (Furthermore, the level of goal attainment, measured with GAS, will also be evaluated at session 6.

Enrolment of people with hand OA will be initiated January 2024. When a maximum of eight people with HOA have been referred for occupational therapy, they will form a group receiving the occupational therapy program. Two groups will receive the occupational therapy program in each municipality. People with HOA referred for occupational therapy, but never completing session1 will be considered as drop-outs. Data will be collected according to the project timeline.

Data analysis Descriptive statistics on ordinal data will be presented with median, range and percentages. Number of people with hand OA refereed and included as well as sessions and components delivered will also be presented. The proportions of people with hand OA with relevant improvement of ADL ability will be presented in the relation to ADL-I, AMPS and goals being reach on the GAS. , Clinically relevant difference/change in the ADL-I is >0.64 logits and clinically relevant change on + 0.3 on the AMPS ADL ability logits has been identified as well as + 0.5 as a statistical relevant change. The levels for goal achievement in the GAS are described in levels from -2 to +2. The participant's current level as "-1, less than expected". The expected goal for the participant under "0, expected level". "+1 and +2, is a description of better or much better than expected" and "-2, is the description of worse than the starting level".

Interviews will be transcribed and analysed to find common patterns in relation to a thematic content analysis related to questions 1, 3, 4, 5.

Ethics The study will be conducted in accordance with the Helsinki declaration and Danish law. Informed consent will be obtained from each participant, including people with hand OA, GPs, and OTs, emphasising the right to withdraw from the study at any time. A copy of the consent form will be provided to participants and the first author will be responsible for saving a consent form in the participant's study file. Each participant is given an ID number, with which all data is pseudonymised and only accessed by authorised personnel obliged to secrecy.

To minimise any risk all GPs and OTs will receive training in the procedures of the HANDY program and the delivery will be by educated and experienced personal.

The results of the study will be reported in accessible formats to study participants, decision makers in the participating municipalities, other stakeholders involved in the study, and public in general. Further, results will be published in peer-reviewed journals and presented on national and international conferences.

ELIGIBILITY:
Inclusion Criteria:

People diagnosed with hand OA, > 18 years and motivated to participate in a group program focusing on improvement in ADL task performance

General practitioners (GPs) working in a clinic with agreement with the Danish health insurance receiving patients with all kinds of everyday symptoms and illnesses, who express interest in contributing to development and evaluation of a program for people with hand OA.

Occupational therapists (OTs) working with community-based rehabilitation and with six months of community-based working experience

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-05-03 (Estimated); Study Completion 2024-06-28 (Estimated)

PRIMARY OUTCOMES:
Participant flow | up to 6 months
  Counts of participant flow

SECONDARY OUTCOMES:
Registration forms from GP | up to 6 months
  Registration forms designed for the study concern:
  1. Yes/NO questions in relation to whether the instructions for the needs evaluations and referral were followed
  2. Likert scale 1 to 5 (1= very low degree, 5= very high degree). Questions in relation to relevance of content in need evaluation and referal procedures
Registration forms from OT | up to 6 months
  Registration forms designed for the study concern:
  1. Yes/NO questions in relation to whether the instructions for occupational intervention session were followed.
     If No the OT can ad a comment about reason and how deviation was made
  2. Likert scale 1 to 5 (1= very low degree, 5= very high degree). Questions in relation to the relevance of content in the occupational intervention session
Registration forms from people with hand osteoarthritis | up to 2 months
  Registration forms from people with hand osteoarthritis concerning perception of content and delivery
  Registration forms designed for the study concern:
  1) Likert scale 1 to 5 (1= very low degree, 5= very high degree). Questions to people with hand osteoarthritis in relation to the perception of content in GP and OT sessions
Observation based ADL motor ability | up to 2 months
  Change in observed ADL motor ability, using the Assessment of Motor and Process Skills (AMPS). Raw ordinal scores are converted into linear, interval scale (i.e. infinite scale) measures of ADL motor ability based on Rasch measurement models and reported in logits.
  Higher measures indicate higher ADL motor ability
Observation based ADL process ability | up to 2 months
  Change in observed ADL motor ability, using the Assessment of Motor and Process Skills (AMPS). Raw ordinal scores are converted into linear, interval scale (i.e. infinite scale) measures of ADL process ability based on Rasch measurement models and reported in logits.
  Higher measures indicate higher ADL process ability
Selfreported ADL ability | up to 2 months
  Change in self-reported ADL ability, using the standardised ADL-Interview (ADL-I). Raw ordinal scores are converted into linear, interval scale (i.e. infinite scale) measures of self-reported ADL ability based on Rasch measurement models and reported in logits.
  Higher measures indicate higher self-reported ADL ability

CONTACTS AND LOCATIONS:
Overall Officials: Eva Elisabet Ejlersen Wæhrens, PhD, Principal Investigator — Parker Institute, Copenhagen University Hospital
Locations (1):
- Parker Institute, Frederiksberg, Capital Region, Denmark

REFERENCES:
- [Background] GBD 2021 Low Back Pain Collaborators. Global, regional, and national burden of low back pain, 1990-2020, its attributable risk factors, and projections to 2050: a systematic analysis of the Global Burden of Disease Study 2021. Lancet Rheumatol. 2023 May 22;5(6):e316-e329. doi: 10.1016/S2665-9913(23)00098-X. eCollection 2023 Jun. PMID 37273833
- [Background] Haugen IK, Englund M, Aliabadi P, Niu J, Clancy M, Kvien TK, Felson DT. Prevalence, incidence and progression of hand osteoarthritis in the general population: the Framingham Osteoarthritis Study. Ann Rheum Dis. 2011 Sep;70(9):1581-6. doi: 10.1136/ard.2011.150078. Epub 2011 May 27. PMID 21622766
- [Background] Andersen U; Doessing, A; Gudbergsen, H; Hagelskjaer, V ; Bliddal, H; Waehrens, EE. Indicators of need for Occupational Therapy. Pending publication.
- [Background] Bukhave EB, Huniche L. Activity problems in everyday life--patients' perspectives of hand osteoarthritis: "try imagining what it would be like having no hands". Disabil Rehabil. 2014;36(19):1636-43. doi: 10.3109/09638288.2013.863390. Epub 2013 Dec 6. PMID 24308906
- [Background] Kloppenburg M, Kroon FP, Blanco FJ, Doherty M, Dziedzic KS, Greibrokk E, Haugen IK, Herrero-Beaumont G, Jonsson H, Kjeken I, Maheu E, Ramonda R, Ritt MJ, Smeets W, Smolen JS, Stamm TA, Szekanecz Z, Wittoek R, Carmona L. 2018 update of the EULAR recommendations for the management of hand osteoarthritis. Ann Rheum Dis. 2019 Jan;78(1):16-24. doi: 10.1136/annrheumdis-2018-213826. Epub 2018 Aug 28. PMID 30154087
- [Background] Kolasinski SL, Neogi T, Hochberg MC, Oatis C, Guyatt G, Block J, Callahan L, Copenhaver C, Dodge C, Felson D, Gellar K, Harvey WF, Hawker G, Herzig E, Kwoh CK, Nelson AE, Samuels J, Scanzello C, White D, Wise B, Altman RD, DiRenzo D, Fontanarosa J, Giradi G, Ishimori M, Misra D, Shah AA, Shmagel AK, Thoma LM, Turgunbaev M, Turner AS, Reston J. 2019 American College of Rheumatology/Arthritis Foundation Guideline for the Management of Osteoarthritis of the Hand, Hip, and Knee. Arthritis Care Res (Hoboken). 2020 Feb;72(2):149-162. doi: 10.1002/acr.24131. Epub 2020 Jan 6. PMID 31908149
- [Background] Lykkegaard J, Møller A and GH. Håndartrose blandt +70 årige i Almen Praksis, Denmark. [Hand Osteoarthritis among +70 year olds in General Practice, Denmark] Copenhagen; 2021.
- [Background] Bobos P, Nazari G, Szekeres M, Lalone EA, Ferreira L, MacDermid JC. The effectiveness of joint-protection programs on pain, hand function, and grip strength levels in patients with hand arthritis: A systematic review and meta-analysis. J Hand Ther. 2019 Apr-Jun;32(2):194-211. doi: 10.1016/j.jht.2018.09.012. Epub 2018 Dec 23. PMID 30587434
- [Background] Takata SC, Wade ET, Roll SC. Hand therapy interventions, outcomes, and diagnoses evaluated over the last 10 years: A mapping review linking research to practice. J Hand Ther. 2019 Jan-Mar;32(1):1-9. doi: 10.1016/j.jht.2017.05.018. Epub 2017 Jun 21. PMID 28647322
- [Background] Kjeken I, Smedslund G, Moe RH, Slatkowsky-Christensen B, Uhlig T, Hagen KB. Systematic review of design and effects of splints and exercise programs in hand osteoarthritis. Arthritis Care Res (Hoboken). 2011 Jun;63(6):834-48. doi: 10.1002/acr.20427. PMID 21630479
- [Background] Osteras N, Kjeken I, Smedslund G, Moe RH, Slatkowsky-Christensen B, Uhlig T, Hagen KB. Exercise for hand osteoarthritis. Cochrane Database Syst Rev. 2017 Jan 31;1(1):CD010388. doi: 10.1002/14651858.CD010388.pub2. PMID 28141914
- [Background] Hand C, Law M, McColl MA. Occupational therapy interventions for chronic diseases: a scoping review. Am J Occup Ther. 2011 Jul-Aug;65(4):428-36. doi: 10.5014/ajot.2011.002071. PMID 21834458
- [Background] Steultjens EM, Dekker J, Bouter LM, Leemrijse CJ, van den Ende CH. Evidence of the efficacy of occupational therapy in different conditions: an overview of systematic reviews. Clin Rehabil. 2005 May;19(3):247-54. doi: 10.1191/0269215505cr870oa. PMID 15859525
- [Background] Skivington K, Matthews L, Simpson SA, Craig P, Baird J, Blazeby JM, Boyd KA, Craig N, French DP, McIntosh E, Petticrew M, Rycroft-Malone J, White M, Moore L. A new framework for developing and evaluating complex interventions: update of Medical Research Council guidance. BMJ. 2021 Sep 30;374:n2061. doi: 10.1136/bmj.n2061. PMID 34593508
- [Background] O'Cathain A, Hoddinott P, Lewin S, Thomas KJ, Young B, Adamson J, Jansen YJ, Mills N, Moore G, Donovan JL. Maximising the impact of qualitative research in feasibility studies for randomised controlled trials: guidance for researchers. Pilot Feasibility Stud. 2015 Sep 7;1:32. doi: 10.1186/s40814-015-0026-y. eCollection 2015. PMID 27965810
- [Background] Fisher AG, Marterella A. Powerful practice: a Model for Authentic Occupational Therapy. Fisher AG, Marterella A, editors. Fort Collins, Colorado, USA: CIOTS - Center for innovative OT solutions..; 2019.
- [Background] Waehrens EE, Nielsen KT. ADL-Interview (ADL-I). Klinisk version 1.0 - Introduktion, ADL-I og administration [Clinical version 1.0 - Introduction, ADL-I, and administration]. Copenhagen; 2020.
- [Background] Waehrens EE, Bliddal H, Danneskiold-Samsoe B, Lund H, Fisher AG. Differences between questionnaire- and interview-based measures of activities of daily living (ADL) ability and their association with observed ADL ability in women with rheumatoid arthritis, knee osteoarthritis, and fibromyalgia. Scand J Rheumatol. 2012 Mar;41(2):95-102. doi: 10.3109/03009742.2011.632380. Epub 2012 Jan 30. PMID 22283877
- [Background] Fisher AG, Jones KB. Assessment of motor and process skills : Volume 1: Development, standardization, and administration manual. 7. ed., Re. Fisher AG, Jones KB, editors. Fort Collins, Colo: Three Star Press; 2012.
- [Background] Fisher AG, Jones KB. Assessment of motor and process skills : Volume 2: User Manual. 7. ed. Fisher AG, Jones KB, editors. Fort Collins, Colo: Three Star Press; 2014.
- [Background] Waehrens EE. Measuring quality of occupational performance based on self-report and observation : development and validation of instruments to evaluate ADL task performance. Sweden, Umeå; 2010.
- [Background] Bard-Pondarre R, Villepinte C, Roumenoff F, Lebrault H, Bonnyaud C, Pradeau C, Bensmail D, Isner-Horobeti ME, Krasny-Pacini A. Goal Attainment Scaling in rehabilitation: An educational review providing a comprehensive didactical tool box for implementing Goal Attainment Scaling. J Rehabil Med. 2023 Jun 14;55:jrm6498. doi: 10.2340/jrm.v55.6498. PMID 37317629
- [Derived] Andersen U, Hagelskjaer V, von Bulow C, Gudbergsen H, Bliddal H, Dossing A, Waehrens EE. A multidisciplinary, cross-sectorial management program for people living with hand osteoarthritis (HANDY): protocol for a feasibility study. Pilot Feasibility Stud. 2025 May 15;11(1):68. doi: 10.1186/s40814-025-01653-1. PMID 40375091